CLINICAL TRIAL: NCT06008171
Title: Patient Decision Aid for the Treatment of Actinic Keratosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-3292
Record Dates: First submitted 2023-07-20; First posted 2023-08-23 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Actinic Keratoses; Patient Decision Aid
Keywords: actinic keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Intervention Model Description: Patients with an indication for treatment of field therapy for actinic keratosis will be consulted with patient decision aid or without patient decision aid (conventional)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient Decision Aid (Active Comparator): Consult about treatment options for field-directed therapies for actinic keratosis by the dermatologist, with the use of a Patient Decision Aid.
  Interventions: Other: Patient Decision Aid
- Without Patient Decision Aid (conventional) (No Intervention): Conventional consult about treatment options for field-directed therapies for actinic keratosis by the dermatologist, without the use of a Patient Decision Aid.

INTERVENTIONS:
Other: Patient Decision Aid — A designed tool (by us) that help patients and providers talk and decide together about field-directed treatment options for actinic keratosis.
  Arms: Patient Decision Aid

SUMMARY:
This study evaluates whether a Patient Decision Aid for the field-directed treatment of actinic keratosis has an effect on shared decision making and patient satisfaction.

DETAILED DESCRIPTION:
Actinic keratosis is the most common epithelial precancerous lesion among the Caucasian race. With an increase in prevalence worldwide due to an aging population and rise of ultraviolet exposure actinic keratosis are among the most frequently encountered skin lesions in clinical practice.

There are many therapeutic modalities for the treatment of actinic keratosis, depending on multiple factors such as distribution, characteristics, patient preference, side effects, availability and costs. Treatment options can be divided into: lesion directed therapy en field directed therapy.

A Patient Decision Aid for field-directed therapies for actinic keratosis may attribute to better shared-decision making and patient satisfaction which on their part may benefits treatment compliance and health outcomes and may lead to fewer disputes between patients and doctors.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis actinic keratosis in MaastrichtUMC+ or CatharinaHospital, Eindhoven
* age >18 years

Exclusion Criteria:

* no knowledge of Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Difference in patient satisfaction | First questionnaire at moment of consultation, between November 2022 and January 2024 (expected). Second questionnaire after finishing the treatment (1 week after consultation up to 6 months after consultation).
  Difference in patient satisfaction making in the group with Patient Decision Aid and the group without Patient Decision Aid, measured with Decision Evaluation Scales.
  This scale uses 15 questions with a maximum score of 75. Higher scores mean more satisfaction and less insecurity.
Difference in shared decision making | First questionnaire at moment of consultation, between November 2022 and January 2024 (expected). Second questionnaire after finishing the treatment (1 week after consultation up to 6 months after consultation).
  Difference in shared decision making in the group with Patient Decision Aid and the group without Patient Decision Aid, measured with Shared Decision Making-Q-9 questionnaire Dutch version.
  This scale uses 9 questions with a maximum score of 45. 0 indicating the lowest and 45 indicating the highest level of perceived shared decision making.

CONTACTS AND LOCATIONS:
Overall Officials: Klara Mosterd, prof.dr., Principal Investigator — Maastricht UMC
Locations (1):
- Ellen Oyen, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No